CLINICAL TRIAL: NCT03476213
Title: Reduction of Awareness and Dreaming During Neurosurgical Procedures Using Target- Controlled Infusion, Comparison With Manual Total Intravenous Anesthesia TIVA.
Brief Title: Manual Versus Targer-controll Infusion in Reduction of Awareness and Dreaming
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Hradec Kralove (Other)
Responsible Party: Principal Investigator, Dostalova Vlasta, MD, PhD, Principal Investigator, University Hospital Hradec Kralove
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 201506S
Record Dates: First submitted 2018-03-09; First posted 2018-03-23 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Anesthesia Awareness
Keywords: Anesthesia Awareness; Dreaming in anesthesia; Total intravenous anesthesia; Target-controll infusion
MeSH Terms: conditions — Intraoperative Awareness

STUDY DESIGN:
Intervention Model Description: Group A will be anesthetized using TIVA, group B using TCI
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group TCI (Experimental): induction and anesthesia will be held by using target-controll infusion
  Interventions: Procedure: Group TCI
- Group TIVA (Active Comparator): induction and anesthesia will be held by manual dosing of propofol and sufentanil
  Interventions: Procedure: Group TIVA

INTERVENTIONS:
Procedure: Group TCI — Induction and anesthesia will be done by using Gepth model for sufentanil and Schnider effect model for propofol. Anesthetics will be aplicated using infusion pump Agilia (Fresenius Kabi). Another titration will be according to target value of entropy between 40 and 60 and surgical pleth index below 35.
  Arms: Group TCI
Procedure: Group TIVA — Induction of anesthesia will be done by titrating of propofol to the dose of 1.2 mg/kg and sufentanil 5-10 ug according to body weight, maintaining of anesthesia using continuous infusion of propofol 5 mg/ kg/hour and sufentanil 35 ug/hour to reach the target value of entropy between 40 and 60 and surgical pleth index below 35.
  Arms: Group TIVA

SUMMARY:
This study compares manual total intravenous anesthesia (TIVA) and target-controll infusion (TCI) in reduction of awareness and dreaming, and the haemodynamical stability during operation. Half of patients will be anesthetized using manual TIVA and other half using TCI.

DETAILED DESCRIPTION:
Awareness is possible in TIVA in case of technical failure or prolonged induction phase, TCI technology seems to prevent these events. Total of 80 patients planed for elective neurosurgical brain tumor resection fulfilling the inclusion criteria will be devided into two groups. First half will be anesthetized using TIVA with manual induction and the second half will be anesthetized using TCI. All patients will fulfil Modified Brice Questionnaire one hour after the end of operation.

ELIGIBILITY:
Inclusion Criteria:

* Glasgow Coma scale 15
* ASA Physical Status Classification System I - III
* planed surgery for brain tumor to 5 hours
* postoperative awakening

Exclusion Criteria:

* NYHA III, IV
* abuse of stimulating drugs, grass, alcohol dependence
* BMI over 40 in females and over 35 in men
* propofol alergie
* awake operations
* postoperative arteficial ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-03-16 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
reduction of awareness | 5 hours
  consciousness during operation

SECONDARY OUTCOMES:
reduction of haemodynamical instability | 5 hours
  reduction of blood pressure by 25 %
reduction of norepinephrine dose | 5 hours
  reduction in ugs during the whole operation

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Dostal, MD, Ph.D., Study Director — University Hospital Hradec Kralove
Locations (1):
- University Hospital Hradec Kralove, Hradec Králové, Czechia